CLINICAL TRIAL: NCT02769832
Title: Phase II Study of Nab-Paclitaxel With Gemcitabine for Relapsed Small Cell Cancer or Those With Progression on First Line Therapy
Brief Title: Nab-Paclitaxel With Gemcitabine for Relapsed Small Cell Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Muhammad Furqan (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor-Investigator, Muhammad Furqan, Clinical Assistant Professor Hematology/Oncology, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201512799
Record Dates: First submitted 2016-01-20; First posted 2016-05-12 (Estimated); Results first posted 2023-07-21 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Small Cell Lung Cancer (SCLC)
Keywords: Abraxane; Albumin-bound Paclitaxel; SCLC; Gemzar
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nab-Paclitaxel with Gemcitabine (Experimental): Nab-paclitaxel 100 mg/m2, day 1 and day 8 of a 21-day cycle Gemcitabine 1000 mg/m2, day 1 and day 8 of a 21-day cycle
  Interventions: Drug: Nab-paclitaxel; Drug: Gemcitabine

INTERVENTIONS:
Drug: Nab-paclitaxel — Nab-paclitaxel 100 mg/m2, day 1 and day 8 of a 21-day cycle
  Other Names: albumin-bound paclitaxel; paclitaxel protein-bound particles for injectable suspension (albumin-bound); Nab-paclitaxel Brand name: Abraxane ®
Drug: Gemcitabine — Gemcitabine 1000 mg/m2, day 1 and day 8 of a 21-day cycle
  Other Names: Generic name: gemcitabine; Brand name: Gemzar ®

SUMMARY:
The purpose of this research study is to see if Abraxane and Gemcitabine given together will be effective in treating small cell cancer that has progressed after one line of treatment.

DETAILED DESCRIPTION:
This study is designed as a second-line therapy for patients with histologically or cytologically confirmed small cell lung cancer or small cell cancer from other organs or poorly differentiated neuroendocrine tumors that are treated like small cell cancer. This study is for patients with metastatic or recurrent disease. Eligible patients will receive Nab-Paclitaxel (Abraxane), 100 mg/m2, IV over 30 minutes on Days 1 and 8 of a 21-day cycle followed by Gemcitabine, 1000 mg/m2, IV over 30 minutes on Days 1 and 8 of a 21-day cycle. Participants can continue receiving Nab-Paclitaxel and Gemcitabine until disease progression, unacceptable toxicity or withdrawal from the study. Tumor measurements will be done every 2 cycles.

ELIGIBILITY:
Inclusion criteria

1. Age ≥18 years old, both male and female
2. Histologically or cytologically confirmed SCLC SCLC or small cell cancer from other organs or poorly differentiated neuroendocrine tumors that are treated like small cell cancer. This study is for patients with metastatic or recurrent disease.
3. ECOG performance status 0-2
4. Patients must have at least one measurable lesion as defined per RECIST 1.1
5. Progression during or after prior first line chemotherapy. Prior maintenance therapy, targeted therapy and immunotherapy are allowed. Prior use of Rovalpituzumab or other ADC agent is allowed. Immunotherapy or targeted therapy if used as 2nd line therapy will not be considered as second line therapy as these are not true chemotherapeutic agents. Patients treated with definitive chemo-radiation will be eligible if they progressed within a year of definitive therapy (as definitive therapy will be considered 1st line therapy for these patients).
6. Before study therapy, a minimum of 21 days must have elapsed since any prior chemotherapy and 2 weeks from the last dose of prior targeted or immunotherapy.
7. Prior definitive XRT is allowed if it has been 2 weeks since the end of definitive XRT. For palliative XRT, protocol-specified treatment can begin at minimum 48 hours after completion of radiation. Lesions within the XRT field can only be used as target lesions if definite progression has been demonstrated since the completion of radiation.
8. Adequate major organ function including the following:

   * Hematologic function: Absolute neutrophil count (ANC) ≥ 1800 /mm3, platelet count ≥ 100,000/mm3, and Hgb ≥ 9.0 gm/dl.
   * Hepatic function: bilirubin ≤ 1.5 x ULN, AST and ALT levels ≤ 2.5 x ULN. If liver metastases are present, then AST and ALT ≤ 5 x ULN.
   * Renal function: serum creatinine ≤ 1.5 x ULN.
9. Patients must be willing and able to sign informed consent for themselves
10. If female: childbearing potential either terminated by surgery, radiation, or menopause, or attenuated by use of an approved contraceptive method (intrauterine device [IUD], birth control pills, or barrier device) during and for 6 months after trial. If male, use of an approved contraceptive method during the study and 6 months afterwards. Females with childbearing potential must have a urine negative hCG test within 7 days prior to the study therapy.

    Females of child-bearing potential (defined as a sexually mature woman who (1) has not undergone hysterectomy [the surgical removal of the uterus] or bilateral oophorectomy [the surgical removal of both ovaries] or (2) has not been naturally postmenopausal for at least 24 consecutive months [i.e., has had menses at any time during the preceding 24 consecutive months]) must:

    Either commit to true abstinence* from heterosexual contact (which must be reviewed on a monthly basis), or agree to use, and be able to comply with, effective contraception without interruption, 28 days prior to starting IP therapy (including dose interruptions), and while on study medication or for a longer period if required by local regulations following the last dose of IP; and

    Have a negative serum pregnancy test (β -hCG) result at screening and agree to ongoing pregnancy testing during the course of the study, as per clinical judgement of the investigator, and after the end of study therapy. This applies even if the subject practices true abstinence* from heterosexual contact.
11. Male subjects must practice true abstinence* or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions and for 6 months following IP discontinuation, even if he has undergone a successful vasectomy.

    * True abstinence is acceptable when this is in line with the preferred and usual lifestyle of the subject. [Periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception].

Exclusion criteria

1. Any of the following because this study involves an agent that has known genotoxic, mutagenic, and teratogenic effects:

   * Pregnant women
   * Nursing women
   * Men or women of childbearing potential, who are unwilling to employ adequate contraception as determined by treating physician, while on this study and for 6 months after the end of treatment with the study drugs.
2. History of the following within the prior 6 months: a myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, New York Heart Association (NYHA) Class III-IV heart failure, uncontrolled hypertension, clinically significant cardiac dysrhythmia or clinically significant ECG abnormality, cerebrovascular accident, transient ischemic attack, or seizure disorder
3. Serious concurrent infection or nonmalignant illness that is uncontrolled or whose control may be jeopardized by complication of study therapy
4. History of other invasive malignancy that is currently active and/or has been treated within 12 months prior to enrollment (notable exceptions include: basal cell carcinoma, squamous cell carcinoma of the skin, localized prostate cancer, in situe carcinomas of the cervix and breast, and superficial bladder cancers [non-muscle invasive]).
5. Psychiatric disorder which, per treating physician discretion, may preclude compliance
6. Major surgery in the last two weeks of starting study therapy. This does not include procedures like biopsy (needle or excisional) or port placement as these are not considered as major surgery.
7. Individuals with the presence of symptomatic CNS metastasis requiring radiation, surgery, or ongoing use of corticosteroids. Untreated or brain metastasis causing any symptoms. Treated brain metastasis must be stable for 4 weeks prior to first dose of study drug and not require steroids for at least 7 days prior to study treatment.
8. Pre-existing peripheral neuropathy > Grade 1 (using CTCAE v 4.3 criteria)
9. Received any prior treatment with any taxane (docetaxel or paclitaxel) for small cell lung cancer.
10. History of allergy or hypersensitivity to albumin-bound paclitaxel, or gemcitabine.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-08-29 (Actual); Primary Completion 2021-09-23 (Actual); Study Completion 2022-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Muhhamad Furqan, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Byrne MM, Sutamtewagul G, Zeitler W, Mott SL, Zamba GKD, Kojadinovic A, Zhang J, Abu-Hejleh T, Clamon G, Furqan M. Phase II study of nab-paclitaxel with gemcitabine for relapsed/refractory small cell lung cancer. Front Oncol. 2024 Jul 31;14:1303268. doi: 10.3389/fonc.2024.1303268. eCollection 2024. PMID 39144826

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Treatment began following screening and within 14 days after screening, if patient is eligible and completed all required testing including medical history, physical exam including performance status, blood samples, pregnancy test, and tumor assessment done by computerized tomography (CT) scan, Chest X-Ray (CXR), or Magnetic Resonance Imaging (MRI).
Groups:
- Nab-Paclitaxel With Gemcitabine: Nab-paclitaxel: 100 mg/m2, day 1 and day 8 of a 21-day cycle; Gemcitabine: 1000 mg/m2, day 1 and day 8 of a 21-day cycle
Period: Overall Study
Arm/Group | Nab-Paclitaxel With Gemcitabine
Started | 32
Completed | 2
Not Completed | 30
Not completed — Death | 30

BASELINE CHARACTERISTICS:
Groups:
- Nab-Paclitaxel With Gemcitabine: Nab-paclitaxel 100 mg/m2, day 1 and day 8 of a 21-day cycle; Gemcitabine 1000 mg/m2, day 1 and day 8 of a 21-day cycle
Arm/Group | Nab-Paclitaxel With Gemcitabine
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 16
Age, Continuous [Mean (Full Range); unit: years] | 64 [48 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 32
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 32
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Overall response rate is defined as the percentage of patients with a confirmed complete or partial response per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI/CT scan:
  Complete response (CR) is the disappearance of all target lesions. Partial Response (PR), is at least a ≥ 30% decrease in the sum of the LD of target lesions taking as reference the baseline sum of the longest diameter (LD). Progression of disease (PD) is at least a ≥ 20% increase in the sum of LD of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions and as defined by RECIST v1.1 guidelines. Stable disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as references the smallest sum LD.
Time Frame: Patients will be evaluated every 2 cycles until progression or off treatment (up to 3 years)
Measure: Count of Participants; unit: Participants
Arm/Group | Nab-Paclitaxel With Gemcitabine
Number analyzed (Participants) | 32
Participants
  Complete Response | 0
  Partial Response | 9
  Stable Disease | 16
  Progressive Disease | 7

2. Secondary Outcome: Progression-Free Survival
Description: Progression-free survival is defined as the time from treatment initiation to the date of first documentation of disease progression or death due to any cause. Otherwise, patients are censored at the date of last radiographic assessment for progression.
Time Frame: Patients will be evaluated every 2 cycles until progression or off treatment (up to 3 years)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nab-Paclitaxel With Gemcitabine
Number analyzed (Participants) | 32
months | 2.9 [2.4 to 3.6]

3. Secondary Outcome: Time to Progression
Description: Time to progression is defined as the time from treatment initiation to the date of first documentation of disease progression per RECIST v1.1. Otherwise, patients are censored at last radiographic assessment for progression.
Time Frame: Patients will be evaluated every 2 cycles until progression or off treatment (up to 3 years)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nab-Paclitaxel With Gemcitabine
Number analyzed (Participants) | 32
months | 2.9 [2.4 to 3.8]

4. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from treatment initiation to death due to any cause. Patients still alive are censored at last date known to be alive.
Time Frame: Patients will be evaluated every 3 months until death or study completion (up to 3 years)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nab-Paclitaxel With Gemcitabine
Number analyzed (Participants) | 32
months | 9.3 [5.2 to 12.4]

ADVERSE EVENTS:
Time Frame: All adverse events were recorded from the time the subject signs informed consent until 28 days after the last dose of Abraxane and Gemcitabine, up to 4 years.
Arm/Group | Nab-Paclitaxel With Gemcitabine
All-Cause Mortality (participants affected / at risk) | 31/32
Serious Adverse Events (participants affected / at risk) | 14/32
Other Adverse Events (participants affected / at risk) | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nab-Paclitaxel With Gemcitabine (N=32)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Duodenal hemorrhage (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Platelet count decreased (Investigations) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Stroke (Nervous system disorders) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitits (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Superior vena cava syndrome (Vascular disorders) | 1 (2)
Thromboembolic event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nab-Paclitaxel With Gemcitabine (N=32)
Anemia (Blood and lymphatic system disorders) | 19 (59)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Heart failure (Cardiac disorders) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (2)
Eye disorders - Other, specify (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (4)
Constipation (Gastrointestinal disorders) | 8 (9)
Diarrhea (Gastrointestinal disorders) | 11 (12)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 5 (6)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 4 (4)
Mucositis oral (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 12 (23)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 8 (18)
Chills (General disorders) | 2 (2)
Edema limbs (General disorders) | 10 (13)
Fatigue (General disorders) | 20 (42)
Fever (General disorders) | 6 (13)
Gait disturbance (General disorders) | 1 (1)
Infusion related reaction (General disorders) | 1 (1)
Infusion site extravasation (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2)
Pain (General disorders) | 1 (1)
Immune system disorders - Other, specify (Immune system disorders) | 1 (1)
Bronchial infection (Infections and infestations) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 2 (2)
Lung infection (Infections and infestations) | 1 (1)
Otitis externa (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 2 (4)
Skin infection (Infections and infestations) | 2 (2)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (5)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 2 (2)
Alanine aminotransferase increased (Investigations) | 3 (8)
Alkaline phosphatase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 4 (6)
Blood bilirubin increased (Investigations) | 1 (2)
Creatinine increased (Investigations) | 3 (3)
GGT increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 22 (46)
Platelet count decreased (Investigations) | 19 (57)
Weight gain (Investigations) | 1 (2)
Weight loss (Investigations) | 7 (14)
Anorexia (Metabolism and nutrition disorders) | 8 (10)
Dehydration (Metabolism and nutrition disorders) | 4 (4)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (6)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 8 (15)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 6 (13)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4)
Cognitive disturbance (Nervous system disorders) | 1 (3)
Dizziness (Nervous system disorders) | 2 (2)
Dysarthria (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (2)
Headache (Nervous system disorders) | 1 (2)
Lethargy (Nervous system disorders) | 1 (1)
Nervous system disorders - Other, specify (Nervous system disorders) | 2 (2)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (5)
Seizure (Nervous system disorders) | 1 (1)
Stroke (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (2)
Insomnia (Psychiatric disorders) | 2 (2)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Nail loss (Skin and subcutaneous tissue disorders) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (4)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 3 (3)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 4 (9)
Phlebitis (Vascular disorders) | 1 (2)
Superior vena cava syndrome (Vascular disorders) | 1 (2)
Thromboembolic event (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-06-23): https://cdn.clinicaltrials.gov/large-docs/32/NCT02769832/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-07): https://cdn.clinicaltrials.gov/large-docs/32/NCT02769832/ICF_001.pdf